CLINICAL TRIAL: NCT07023692
Title: Visual and Auditory Distraction for the Relief of Pain and Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-02133-01
Record Dates: First submitted 2025-04-15; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Bone Marrow Aspiration; Pain; Anxiety; Hematologic Diseases; Hematologic Disorders; Visual Distraction; Auditory Distraction
Keywords: pain perception; anxiety; nociceptive response; relief of pain; relief of anxiety; visual distraction; auditory distraction
MeSH Terms: conditions — Pain; Anxiety Disorders; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Distraction with VR headsets during bone marrow examinations
  Interventions: Behavioral: Distraction with VR (Virtual Reality) headsets
- Control group (No Intervention): Bone marrow examinations according to standard procedure

INTERVENTIONS:
Behavioral: Distraction with VR (Virtual Reality) headsets — VR headsets will be fitted and applied in consultation with the study participants. Distraction material will be selected from a range of options based on the participant's preferences, such as watching/listening to a story, an experience of being in nature, or mindfulness. When applying the VR headsets, care will be taken to ensure no light leaks into the eyes and that the headband and headphones are not perceived as too tight. This is especially important in terms of the risk for motion sickness (cyber sickness). The VR headsets will then be used throughout the examination procedure and removed once the bandage has been applied.
  Arms: Intervention group

SUMMARY:
Bone marrow (BM) examinations are performed in diagnostic workup of malignancies, in particular hematological diseases, and are frequently associated with significant pain, distress, and anxiety. Analgesic and sedative medications are given to alleviate discomfort.

The aim of this project is to study the effects of visual and auditory distraction on pain and anxiety during BM examinations.

The project includes two baseline studies assessing pain perception, anxiety, and nociceptive response in patients and healthy volunteers undergoing BM examinations, and two randomized controlled trials evaluating the efficacy of VR distraction in reducing pain perception, anxiety, and nociceptive response. The intervention groups will use VR headsets, while control groups will follow standard procedure. Data collection include measurements of skin conductance, pulse, validated questionnaires and qualitative interviews.

The project is strongly anchored in clinical practices and is a collaboration between Skåne University Hospital and Lund University, Sweden. The project group consists of three experts with relevant clinical and research competences. The project is ongoing, data collection will be finalized in 2028, and analyses and publications in 2027-2029.

If distraction with VR results in less painful examinations and shows to be feasible in clinical praxis, the findings may contribute to development of new guidelines for pain management in BM-examinations and other painful medical procedures.

DETAILED DESCRIPTION:
Purpose and aims: The overall aim of this project is to study the effect of visual and auditory distraction as a relief for pain and anxiety in adults undergoing bone marrow aspiration and/or biopsy. The goal is to increase knowledge about pain and pain relief during bone marrow procedures, as well as to explore whether there is a difference in pain responses and experiences of health, anxiety, and pain between patients and healthy volunteers. Additionally, the project aims to investigate whether individuals undergoing bone marrow examinations can experience less anxiety and pain compared to standard procedures through visual and auditory distraction via VR, and whether pain relief can be made more individualized and person centered.

Specific objectives:

To evaluate if it is possible to measure anxiety-induced stress responses and pain in individuals undergoing bone marrow examinations during standard procedures with objective measurement tools (skin conductance and pulse).

To evaluate how individuals rate their health, anxiety, and pain after a bone marrow examination.

To evaluate if there is a difference in anxiety-induced stress responses and pain between patients and healthy volunteers undergoing bone marrow examinations with VR versus without VR.

To evaluate if there is a difference in self-reported health, anxiety, and pain between patients and healthy volunteers undergoing bone marrow examinations with VR versus without VR.

To evaluate if there is a difference in patients' and healthy volunteers' experiences of a bone marrow examination with VR versus without VR.

To evaluate if there is a difference in the dosage of local anesthetics and any sedative medications used during a bone marrow examination with VR versus without VR.

To evaluate the staff's perceptions of the approach to bone marrow examinations with VR versus without VR.

State-of-the art: Bone marrow examinations are conducted for the diagnosis and follow-up of various hematological diseases and treatments. The purpose is to search for, confirm, or exclude a hematological diagnosis, or to evaluate the effectiveness of treatment for an already established disease. The majority of patients with hematological diseases typically undergo several bone marrow examinations during their disease and treatment periods.

Bone marrow samples are typically taken from the back of the hip bone. To optimize the placement of the sampling site, the patient is usually positioned on their side with knees drawn up and bent. Local anesthesia is commonly used for adults undergoing bone marrow examinations, while general anesthesia is rarely used, whereas it is routine for children (<18 years old). The bone marrow sample is taken using a relatively large needle that is inserted through the skin and approximately half a centimeter into the hip bone, where a small amount of bone marrow is aspirated, alternatively, a tissue sample of the bone marrow is taken. Bone marrow examinations usually take about 15-20 minutes.

For the patient, bone marrow examinations are often perceived as a painful and uncomfortable experience, and are therefore frequently associated with anxiety, which is often related to concerns about the results of the examination. Various pain relief regimens are used, with Lidocaine-based local anesthesia being the most common. However, there are no clear guidelines regarding the anesthesia procedure for bone marrow examinations.

A few studies have been conducted to investigate the effect of VR headsets as a form of reality diversion on pain and anxiety during bone marrow examinations, which indicate that VR headsets are well-tolerated and that patients, nurses, and physicians report satisfaction. However, the effect of VR headsets on pain intensity has shown varying results, suggesting that more studies are needed. In previous studies, pain and anxiety have been measured using self-report tools, but without objective measurements of pain.

Objective measurements of pain response (nociception) are currently available both in research and commercially through a variety of techniques. One of the most common and well-studied methods is the Nociception Level Index (NOL) from Medasense, which uses a fingertip sensor to measure physiological values and then presents the degree of nociception numerically. Additionally, the PainSensor from MedStorm (PAM), a sensor attached to the palm of the hand, measures changes in the skin's ability to conduct electrical signals (skin conductance) and provides a nociception value based on this.

Using VR headsets means that the patient wears glasses and headphones that place them in a virtual reality while still being able to communicate with the responsible staff. The examination can thus be tailored to the individual as well as designed in a way that hopefully provides the patient with enhanced experience and better pain relief outcomes. Currently, VR is not routinely used as a distraction during bone marrow examinations. The goal is that this research project will lead to increased patient satisfaction regarding perceived pain and anxiety, as well as involvement in decision-making about pain relief methods, and that additional knowledge about the procedure will be gained.

Significance and scientific novelty: The use of VR for distraction is rare in clinical practice. The originality of this project primarily lies in its strong clinical foundation, which allows for direct implementation of the results into clinical practice. This could potentially benefit patients in the near future after the project's conclusion. The project is rooted in clinical practice, utilizing VR in conjunction with bone marrow examinations. Bone marrow examinations are necessary and recurring for patients with hematological diagnoses, most often cancer, for the selection of further treatments, and are crucial for the patient's diagnosis, disease status, and prognosis. Having a hematological diagnosis means undergoing multiple treatments over an extended period, which involves many hospitalizations with demanding treatments, discomfort, illness, and pain. Distraction with VR could make these examinations feel less stressful, potentially making the patient's pain more tolerable and reducing time spent in the hospital during the examinations, as well reducing the use of opioids and their troublesome side effects.

Preliminary and previous results: The development phase of the project, including a Proof of Concept (POC) study, was conducted in the spring of 2024. The concept was tested on eight patients who underwent bone marrow examinations according to the standard procedure, all of whom had prior experience with this examination, and demonstrated good feasibility. At the end of the autumn of 2024, the project started with the first study, which involves measuring nociceptive responses using conductance monitoring and pulse during bone marrow examinations according to the standard procedure, as well as administering questionnaires to patients and staff after the examination.

Project description, Theory and method:

The project is designed as a complex intervention study and consists of four studies: two observational studies (baseline) with patients (Study 1) and healthy volunteers (Study 2) undergoing bone marrow examination according to the standard procedure, and two randomized intervention studies with patients (Study 3) and healthy volunteers (Study 4) undergoing bone marrow examination in two arms:

The intervention group: Distraction with VR headsets during bone marrow examinations The control group: Bone marrow examinations according to standard procedure

The total number of participants expected to be included is approximately 220 patients and 40-80 healthy volunteers:

Data collection:

During the ongoing bone marrow examination: In all four studies, objective markers measuring the level of pain (nociception) will be studied. Nociceptive response will be monitored using the two techniques NOL and MedStorm PainSensor, as well as pulse recordings using an additional finger clamp.

Immediately after the bone marrow examination:

In all four studies, questionnaires will be given to the study participants (patients and healthy volunteers) with questions regarding demographics (age and gender), the number of previous bone marrow examinations, and any ongoing pain and/or anxiety issues, including the location of any pain. Additionally, validated self-reported instruments will be used.

Individual interviews with approximately 20 patients (Study 3) and around 10 healthy volunteers (Study 4) will be conducted to gain deeper insight into their experiences with the use of VR headsets, their sense of involvement, pain, and anxiety. Individual interviews will also be carried out with about 10 staff members who have been involved in bone marrow examinations where VR headsets were used, to gather in-depth knowledge about their experiences.

Time plan and implementation:

Ethical approval from the Ethics Review Authority (EPM) was obtained on June 17, 2024, Dnr 2024-02133-01.

Proof of Concept (POC) was conducted in the spring of 2024, which demonstrated good feasibility.

The project was planned and initiated in the fall of 2024. The inclusion and implementation of Study 1 began toward the end of 2024 and is ongoing, with completion expected in June 2026. Study 2 is being conducted in parallel.

Data analysis from Studies 1 and 2 are scheduled for the fall of 2026, with results expected to be ready for publication in 2027.

Studies 3 and 4 are planned to take place in 2027 - 2028, with analysis in 2028 and publication ready by 2029.

The project is expected to conclude in 2029, with clinical implementation planned post-2029, including the dissemination of the intervention to other centers conducting bone marrow biopsies.

Project organization:

The project is carried out in collaboration between the Department of Hematology, Oncology, and Radiation Physics at Skåne University Hospital (SUS) and the Department of Health Sciences (IHV), Faculty of Medicine, Lund University (LU). The project group consists of experts with relevant clinical and research competencies. The members of the project group have extensive experience working with all the scientific approaches involved in the project, ensuring the execution and credibility of the results.

Baseline studies are ongoing. Power analysis will be performed in a post baseline using the Power and Sample Size Program prior to the intervention study. However, previous literature indicates that the number of patients for a randomized study should be at least n = 100. Regarding the risk of non-response, we should increase the number of people included in the study by 10%, which means including a total of 110 study patients, 55 per group: intervention and control.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients
* Adult (≥18 years) healthy volunteers without a hematological diagnosis undergoing bone marrow examination (aspiration and/or biopsy) at the Hematology Out-Patient Care Unit at SUS in Lund, Sweden.

Exclusion Criteria:

* Individuals who cannot understand information and instructions
* Pregnant women
* Persons with skin injuries at the bone marrow examination site
* Those unable to lie on their side
* hearing and/or severe vision impairment
* those prone to motion sickness
* participation in the study during a previous bone marrow examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Nociceptive response | Periprocedural
  Objective markers measuring the level of pain, nociceptive response, monitored by using the the NOL technique, which presents an indexed value between 0 and 100 (i.e. units on a scale), where a higher score means worse outcome, i.e., higher nociceptive response.
Nociceptive response | Periprocedural
  Objective markers measuring the level of pain, nociceptive response, monitored by using the the MedStorm PainSensor technique, which presents an indexed value between 0 and 10 (i.e. units on a scale), where a higher score means worse outcome, i.e., higher nociceptive response.
Self-reported subjective health | Immediately after the bone marrow examination - Periprocedural
  Questionnaires will be given to the study participants with validated self-reported instrument Perceived Health: RAND-36 - RAND Corporation (Research and Development), reporting a score, 0 - 100 points on a scale, where a higher score means better outcome, i.e. the better health.
Self-reported subjective pain | Immediately after the bone marrow examination - Periprocedural
  Questionnaires will be given to the study participants with the validated self-reported instrument Self-reported Pain: NRS - Numerical Rating Scale, where pain is indicated on a scale of 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Self-reported subjective anxiety | Immediately after the bone marrow examination - Periprocedural
  Questionnaires will be given to the study participants with the validated self-reported instrument Self-reported Anxiety: STAI - State-Trait Anxiety Inventory. A score will be reported on a scale, where the scores range between 20-80 points, where a higher score means worse outcome, i.e., higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Heart rate | Periprocedural
  Pulse recordings using an additional finger clamp

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Out-Patient Care Unit , Department of hematology, oncology and radian physics, Skåne University Hospital (SUS) in Lund, Sweden, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not of any value to be shared since the focus is to gather data on a group level.

REFERENCES:
- [Background] Jildenstal P, H.K., Almskog K, et al., Monitoring the Nociception Level Intraoperatively - An Initial Experiences. J Anest & Inten Care, 2018. Med. 7(2): p. 555709.
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Hays RD, Morales LS. The RAND-36 measure of health-related quality of life. Ann Med. 2001 Jul;33(5):350-7. doi: 10.3109/07853890109002089. PMID 11491194
- [Background] Karsh BT. Beyond usability: designing effective technology implementation systems to promote patient safety. Qual Saf Health Care. 2004 Oct;13(5):388-94. doi: 10.1136/qhc.13.5.388. PMID 15465944
- [Background] Rycroft-Malone J. The PARIHS framework--a framework for guiding the implementation of evidence-based practice. J Nurs Care Qual. 2004 Oct-Dec;19(4):297-304. doi: 10.1097/00001786-200410000-00002. No abstract available. PMID 15535533
- [Background] Norbeck DW, Lindgren S, Wolf A, Jildenstal P. Reliability of nociceptive monitors vs. standard practice during general anesthesia: a prospective observational study. BMC Anesthesiol. 2025 Jan 31;25(1):51. doi: 10.1186/s12871-025-02923-4. PMID 39891061
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Spielberger CD, Vagg PR. Psychometric properties of the STAI: a reply to Ramanaiah, Franzen, and Schill. J Pers Assess. 1984 Feb;48(1):95-7. doi: 10.1207/s15327752jpa4801_16. No abstract available. PMID 6707862
- [Background] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Hoffman HG, Richards TL, Van Oostrom T, Coda BA, Jensen MP, Blough DK, Sharar SR. The analgesic effects of opioids and immersive virtual reality distraction: evidence from subjective and functional brain imaging assessments. Anesth Analg. 2007 Dec;105(6):1776-83, table of contents. doi: 10.1213/01.ane.0000270205.45146.db. PMID 18042882
- [Background] Soret L, Gendron N, Rivet N, Chocron R, Macraigne L, Clausse D, Cholley B, Gaussem P, Smadja DM, Darnige L. Pain Assessment Using Virtual Reality Facemask During Bone Marrow Aspiration: Prospective Study Including Propensity-Matched Analysis. JMIR Serious Games. 2022 Oct 12;10(4):e33221. doi: 10.2196/33221. PMID 36222814
- [Background] Le Du K, Septans AL, Maloisel F, Vanquaethem H, Schmitt A, Le Goff M, Clavert A, Zinger M, Bourgeois H, Dupuis O, Denis F, Bouchard S. A New Option for Pain Prevention Using a Therapeutic Virtual Reality Solution for Bone Marrow Biopsy (REVEH Trial): Open-Label, Randomized, Multicenter, Phase 3 Study. J Med Internet Res. 2023 Feb 15;25:e38619. doi: 10.2196/38619. PMID 36790852
- [Background] Korkmaz E, Guler S. The Effect of Video Streaming With Virtual Reality on Anxiety and Pain During Bone Marrow Aspiration and Biopsy Procedure. Pain Manag Nurs. 2023 Dec;24(6):634-640. doi: 10.1016/j.pmn.2023.04.014. Epub 2023 May 27. PMID 37246094
- [Background] Boland JW. Effect of Opioids on Survival in Patients with Cancer. Cancers (Basel). 2022 Nov 21;14(22):5720. doi: 10.3390/cancers14225720. PMID 36428812
- [Background] Bezu L, Rahmani LS, Buggy DJ. The effect of the type of anaesthesia on long-term outcomes after cancer resection surgery: a narrative review. Anaesthesia. 2025 Feb;80(2):179-187. doi: 10.1111/anae.16464. Epub 2025 Jan 8. PMID 39777733
- [Background] Zahid MF. Methods of reducing pain during bone marrow biopsy: a narrative review. Ann Palliat Med. 2015 Oct;4(4):184-93. doi: 10.3978/j.issn.2224-5820.2015.09.02. PMID 26541397
- [Background] Gendron N, Zia Chahabi S, Poenou G, Rivet N, Belleville-Rolland T, Lemaire P, Escuret A, Ciaudo M, Curis E, Gaussem P, Siguret V, Darnige L. Pain assessment and factors influencing pain during bone marrow aspiration: A prospective study. PLoS One. 2019 Aug 29;14(8):e0221534. doi: 10.1371/journal.pone.0221534. eCollection 2019. PMID 31465426
- [Background] Liptrott SJ, Botti S, Bonifazi F, Cioce M, De Cecco V, Pesce AR, Caime A, Rostagno E, Samarani E, Galgano L, Ciceri F, Orlando L, Gargiulo G. Management of Pain and Anxiety during Bone Marrow Aspiration: An Italian National Survey. Pain Manag Nurs. 2021 Jun;22(3):349-355. doi: 10.1016/j.pmn.2020.09.005. Epub 2020 Oct 24. PMID 33109451
- [Background] Bain BJ. Morbidity associated with bone marrow aspiration and trephine biopsy - a review of UK data for 2004. Haematologica. 2006 Sep;91(9):1293-4. PMID 16956842
- [Background] Vanhelleputte P, Nijs K, Delforge M, Evers G, Vanderschueren S. Pain during bone marrow aspiration: prevalence and prevention. J Pain Symptom Manage. 2003 Sep;26(3):860-6. doi: 10.1016/s0885-3924(03)00312-9. PMID 12967736
- [Background] Kuivalainen AM, Pitkaniemi J, Widenius T, Elonen E, Rosenberg P. Anxiety and pain during bone marrow aspiration and biopsy. Scand J Pain. 2012 Apr 1;3(2):92-96. doi: 10.1016/j.sjpain.2011.11.002. PMID 29913774
- [Background] Alzanad F, Feyaza M, Chapanduka ZC. A study of patient-reported pain during bone marrow aspiration and biopsy using local anesthesia alone compared with local anesthesia with intravenous midazolam coadministration at a tertiary academic hospital in South Africa. Health Sci Rep. 2022 Oct 31;5(6):e902. doi: 10.1002/hsr2.902. eCollection 2022 Nov. PMID 36324428
- [Background] Johnson H, Burke D, Plews C, Newell R, Parapia L. Improving the patient's experience of a bone marrow biopsy - an RCT. J Clin Nurs. 2008 Mar;17(6):717-25. doi: 10.1111/j.1365-2702.2007.01991.x. Epub 2007 Nov 30. PMID 18047576
- See also: We have extensive clinical and research networks both nationally and internationally, including groups from Lund University and Gothenburg University with extensive knowledge and experience in pain management. — https://www.gu.se/forskning/malstyrd-icke-invasiv-monitoreringsteknik-under-anestesi